CLINICAL TRIAL: NCT02991404
Title: Single Injection Adductor Canal Block Versus Continuous Adductor Canal Infusion for Total Knee Arthroplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00041950
Record Dates: First submitted 2016-12-08; First posted 2016-12-13 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Total Knee Arthroplasty; Pain, Postoperative; Adductor Canal Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continuous adductor canal block (Active Comparator): After successful placement of the adductor canal catheter placed in standard fashion , the patient will receive a one-time (Initial bolus) 20 ml bolus of 0.25% bupivacaine, 1.67 mcg/ml of clonidine, and 1:400,000 epinephrine followed by a continuous infusion of 0.125% bupivacaine set at 10ml/hour.
  Multimodal peripheral nerve block injection.
  Interventions: Procedure: Multimodal Peripheral Nerve Block Injection; Drug: Initial Bolus; Drug: Continuous infusion
- Single injection block with sham cath (Sham Comparator): Single Shot Adductor Canal Block . Patients will receive single injection adductor canal block (Initial Bolus) with bupivacaine 0.25%, epinephrine, clonidine, buprenorphine and dexamethasone. These patients will have a sham infusion catheter of inert saline placed in the same fashion as the other group.
  Interventions: Procedure: Single Shot Adductor Canal Block; Drug: Initial Bolus

INTERVENTIONS:
Procedure: Multimodal Peripheral Nerve Block Injection — After successful placement of the adductor canal catheter placed in standard fashion , the patient will receive a one-time 20 ml bolus of 0.25% bupivacaine, 1.67 mcg/ml of clonidine, and 1:400,000 epinephrine followed by a continuous infusion of 0.125% bupivacaine set at 10ml/hour.
  Other Names: adductor canal catheter bolus and continuous infusion
  Arms: Continuous adductor canal block
Procedure: Single Shot Adductor Canal Block — A total of 20 ml of solution containing a combination of 0.25% bupivacaine, 1.67 mcg/ml of clonidine, 150 micrograms of buprenorphine, 2 mg of dexamethasone, and 1:400,000 epinephrine will be administered underneath the Sartorius muscle. A sham catheter will then be placed subcutaneously into the Sartorius muscle, secured in typical fashion, and connected to a pump containing saline to provide similar shape and weight with an opaque bag covering the pump. The pump will be run at the lowest possible ml/hour rate, which is currently 0.1 ml/hour with the current pump used in our hospital.
  Other Names: adductor canal block
  Arms: Single injection block with sham cath
Drug: Initial Bolus — 20 ml bolus of 0.25% bupivacaine, 1.67 mcg/ml of clonidine, and 1:400,000 epinephrine
Drug: Continuous infusion — Continuous infusion of 0.125% bupivacaine
  Arms: Continuous adductor canal block

SUMMARY:
Patients undergoing Primary Total Knee Arthroplasty will be randomized to receive either multimodal single injection adductor canal block with sham infusion catheter or continuous infusion of local anesthetic (control) for postoperative analgesia.

Primary end point is pain scores at 30 hours post performance of block procedure.

DETAILED DESCRIPTION:
The objective of this study is to determine if a single shot multimodal peripheral nerve block containing bupivacaine, dexamethasone, buprenorphine, clonidine, and epinephrine will provide comparable (equivalent) analgesic control when compared to an adductor catheter. The primary end point will be pain scores at 30 hours post block initiation. Secondary end points will include, opioid consumption, time to first analgesic request; pain scores; binary patient satisfaction (yes/no); likeliness to recommend their analgesic regimen, straight leg raise test on post-operative day (POD) number 1; adverse events, incidence of post-operative nausea, and vomiting.

Methods and Measures Design The study will be a randomized, double-blind, sham catheter study. Patients will be recruited and randomized to one of two groups: The "Treatment Arm" receive a single shot adductor canal block containing 20 milliliters (ml) of solution including 0.25% bupivacaine, 150 mcg of buprenorphine, 2 mg of dexamethasone, 1.67 mcg/ml of clonidine, and 1:400,000 epinephrine with sham catheter. The sham catheter will be placed in the Sartorius muscle in the same sterile, aseptic fashion as patient's in the control arm. The pump will be set at the lowest possible volume per hour of normal saline (0.1 ml/hour in the current pump in use at our hospital). An opaque bag will be placed over the pump for blinding purposes. The "Control Arm" will receive an adductor canal catheter through which they will receive a 20 ml bolus of 0.25% bupivacaine with 1:400,000 epinephrine followed by an adductor canal catheter infusion of 0.125% bupivacaine at 10 ml/hour. An opaque bag will be placed over the control arm pumps in similar fashion. For all patients, the order in the electronic medical record will be per research pharmacy protocol. For their primary anesthetic, patients in both arms will then receive either a subarachnoid (spinal) anesthetic or general anesthetic per the anesthesiologist in the operating room.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion in the study if they are:

* Age of 18 years old or older
* Scheduled to primary unilateral total knee arthroplasty.
* Patients must give written informed consent for anesthesia including continuous adductor canal block for postoperative analgesia prior to recruitment

Exclusion Criteria:

Patients will be excluded if they have:

* A contraindication to an adductor canal block or catheter placement including, but not limited to site infection, irritation, or refusal.
* Poorly controlled diabetes (A1C >8.0)
* Allergy to medications involves in this study (opioids, bupivacaine, buprenorphine, clonidine, or dexamethasone)
* Opioid use >40 mg of oxycodone daily, long-acting opioids.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Pain scores | 30 hours post block placement
  At 30 hours pain scores between the two groups will be compared for determining statistically significant differences

SECONDARY OUTCOMES:
total opioid consumption | Through 30 hours post block
  The amount of total opioid consumed will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Jaffe, D.O., Principal Investigator — Dr.
Locations (1):
- Wake Forest Baptist Hospital, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No